CLINICAL TRIAL: NCT02262000
Title: A Phase II Clinical Trial of Image Guided Stereotactic Ablative Radiotherapy (SABR) for T2 and Microscopic T3 (PL3), N0,M0 Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Image Guided Stereotactic Ablative Radiotherapy for Non-Small Cell Lung Cancer
Acronym: SABR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: West Virginia University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU010513
Record Dates: First submitted 2014-09-25; First posted 2014-10-10 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Surgically inoperable; Radiation Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - 7.5 Gy x 10 daily fractions (Experimental): Radiotherapy: 7.5 Gy x 10 daily fractions delivered with VMAT or regular IMRT at West Virginia University.
  Interventions: Radiation: Image Guided Stereotactic Ablative Radiotherapy
- B - 12 Gy x 5 daily fractions (Experimental): Radiotherapy: Optional schedule of 12 Gy x 5 daily fractions can may also be used ONLY in situations where dose constraints for organs at risk can be EASILY met while optimal PTV coverage is achieved
  Interventions: Radiation: Image Guided Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Image Guided Stereotactic Ablative Radiotherapy
  Other Names: SABR

SUMMARY:
This study will help researchers learn about the best dose of radiation to be used when treating large early stage non-small cell lung cancer (NSCLC) with a treatment called stereotactic ablative radiotherapy (SABR). Current treatments with SABR for early stage NSCLC show positive response. But, for large early stage NSCLC it may be better to give different SABR doses than what is used in routine early stage NSCLC treatment. It is not understood which dose is best for treating large early stage NSCLC. Therefore, this study can help researchers learn if giving a higher dose using SABR over a period of 5-10 treatment days can increase the chance of cure for large early stage NSCLC.

DETAILED DESCRIPTION:
Treatment Plan:

7.5 Gy x 10 daily fractions delivered with volumetric modulated arc therapy (VMAT) or regular intensity-modulated radiation therapy (IMRT).

* Optional schedule of 12 Gy x 5 daily fractions can may also be used ONLY in situations where dose constraints for organs at risk can be EASILY met while optimal planning target volume (PTV) coverage is achieved; but the 7.5 Gy x 10 daily fractions schedule is preferred.
* All doses are prescribed to the tumor periphery.

For this protocol, patients will be followed only up to 2 years post radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell Lung Cancer
* T2N0M0 or T3(PL3)N0M0 or Locally recurrent ≤ 7 cm
* Surgically inoperable
* ECOG Performance 0-2

Exclusion Criteria:

* Pacemaker on the same side of the tumor
* Pregnant
* Infection that requires IV antibiotics
* Concomitant or adjuvant anti-neoplastic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07-07 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Mattes, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy A, Guckenberger M, Hurkmans C, Nestle U, Belderbos J, De Ruysscher D, Faivre-Finn C, Le Pechoux C. SBRT Dose and Survival in Non-Small Cell Lung Cancer: In Regard to Koshy et al. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):945-6. doi: 10.1016/j.ijrobp.2015.03.032. No abstract available. PMID 26104945

RESULTS

PARTICIPANT FLOW:
Groups:
- A - 7.5 Gy x 10 Daily Fractions: Radiotherapy: 7.5 Gy x 10 daily fractions delivered with volumetric modulated arc therapy (VMAT) or regular intensity-modulated radiation therapy (IMRT) at West Virginia University.
  Image Guided Stereotactic Ablative Radiotherapy
- B - 12 Gy x 5 Daily Fractions: Radiotherapy: Optional schedule of 12 Gy x 5 daily fractions can may also be used ONLY in situations where dose constraints for organs at risk can be EASILY met while optimal planning target volume (PTV) coverage is achieved
  Image Guided Stereotactic Ablative Radiotherapy
Period: Overall Study
Arm/Group | A - 7.5 Gy x 10 Daily Fractions | B - 12 Gy x 5 Daily Fractions
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants from B - 12 Gy x 5 daily fractions were enrolled in the study.
Groups:
- A - 7.5 Gy x 10 Daily Fractions: Radiotherapy: 7.5 Gy x 10 daily fractions delivered with VMAT or regular IMRT at West Virginia University.
  Image Guided Stereotactic Ablative Radiotherapy
- B - 12 Gy x 5 Daily Fractions: Radiotherapy: Optional schedule of 12 Gy x 5 daily fractions can may also be used ONLY in situations where dose constraints for organs at risk can be EASILY met while optimal PTV coverage is achieved
  Image Guided Stereotactic Ablative Radiotherapy
- Total: Total of all reporting groups
Arm/Group | A - 7.5 Gy x 10 Daily Fractions | B - 12 Gy x 5 Daily Fractions | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate (Absence of Local Progression) Using SABR for Treatment of NSCLC
Time Frame: 2 years
Population: Data is not available because the study was terminated and the original PI left the institution. All efforts were made to contact the PI/study team, but we were unsuccessful. No outcome measures data was available.
Arm/Group | A - 7.5 Gy x 10 Daily Fractions | B - 12 Gy x 5 Daily Fractions
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Best Response
Description: To determine the 2-year regional, and distant metastasis rates, progression-free survival (PFS), local progression free survival (L-PFS), overall survival (OS)
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | A - 7.5 Gy x 10 Daily Fractions | B - 12 Gy x 5 Daily Fractions
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Data is not available because the study was terminated and the original PI left the institution. All efforts were made to contact the PI/study team, but we were unsuccessful. No adverse event data was available.
Arm/Group | A - 7.5 Gy x 10 Daily Fractions | B - 12 Gy x 5 Daily Fractions
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes